CLINICAL TRIAL: NCT05952674
Title: Resistant Depression and Vagus Nerve Stimulation : a Medico-economic, Multicenter, Randomized and Open Trial
Brief Title: Treatment Resistant Depression and Vagus Nerve Stimulation
Acronym: DepVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200066
Record Dates: First submitted 2021-05-27; First posted 2023-07-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Treatment Resistant Depression (TRD)
Keywords: Treatment Resistant Depression (TRD); Vagus Nerve Stimulation (VNS); Best Medical Treatment (BMT)
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Patients (166) suffering from resistant depression will be enrolled over a 24-month period and will be randomized in a (1:1) ratio to receive either Vagus Nerve Stimulation (VNS) along with the Best Medical Treatment (VNS+BMT arm) or the Best Medical Treatment only (BMT arm).
Masking Description: None of the parties involved in this research will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus Nerve Stimulation (VNS) + Best Medical Treatment (BMT) (Experimental): Along with the Optimal Medical Treatment for resistant depression, the VNS + BMT arm will be implanted a medical device of VNS.
  Interventions: Device: Vagus Nerve Stimulation (VNS)
- Best Medical Treatment (Active Comparator): The BMT arm will only receive the Optimal Medical Treatment for resistant depression.
  Interventions: Other: Best Medical Treatment

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) — The surgical intervention for the implantation of the VNS medical device is performed by a neurosurgeon under general anesthesia and lasts about an hour. Two incisions are made on the left: one incision to implant an electrode wrapped around the vagus nerve, the other incision to implant the stimulator. The electrode and the stimulator are connected by a cable tunneled. The cardiac tolerance is usually tested at the end of the surgery by turning on the neurostimulator for a few minutes. The stimulator is turned on about two weeks after the implantation, and after the neurosurgeon has checked the quality of healing. The settings used in first intention are standardized and derived from the parameters usually used for the treatment of epilepsies: a pulse width of 250μs, a stimulation frequency of 30Hz, and a 30sec stimulation cycle (ON) every 5min (OFF). Intensity is progressively increased by steps of 0.25mA to reach the 1.5-2mA range, depending on stimulation-induced side effects.
  Arms: Vagus Nerve Stimulation (VNS) + Best Medical Treatment (BMT)
Other: Best Medical Treatment — Best Medical Treatment for resistant depression.
  Arms: Best Medical Treatment

SUMMARY:
Depression is a common illness, affecting 17% of the population over the course of a lifetime. A third of depressions relapses and progresses to recurrence and resistance to treatments. Despite the optimization of antidepressant medical strategies, 20 to 40% of depressions do not respond to treatment. This is particularly worrying as 6% of non-responder patients will die by committing suicide.

Depression has a major impact on quality of life, socio-professional functioning and healthcare consumption.

Sometimes, TRD is part of a bipolar illness. In this case, the challenge is even bigger because antidepressants are no well tolerated, further reducing the therapeutic options in case of resistance, the severity and duration of the depressive episodes are the main factors explaining the deterioration of the quality of life and the increasing cost of cares for these patients.

The standard treatment for TRD is electroconvulsive therapy (ECT), which results in a response in 60 to 70% of cases after a few weeks of treatment. However, the improvement is often transient and 40% of patients relapse within 6 months of the initial ECT session. Moreover, ECT is often not well tolerated. This therapeutic impasse therefore makes TRD a priority public health target to which it is urgent to provide a realistic medico-economical response.

The literature suggests that Vagus Nerve Stimulation (VNS) has unique kinetics of efficacy in depression, particularly in preventing long-term recurrences, and therefore responding to the lack of effective maintenance treatment in TRD. In fact, the benefits of VNS gradually accumulate over 12-24 months, which makes it complementary to more incisive treatments like ECT. Finally, its efficacy-tolerance profile appears to be similar in uni and bipolar TRD, giving VNS a potentially unique place in the therapeutic arsenal in psychiatry.

The DepVNS hypothesis is that VNS is a medico-economically efficient therapeutic option to overcome the therapeutic impasse in which patients suffering from uni and bipolar DR currently find themselves due to the frequency of relapses under treatment.

The primary objective is to estimate, from a collective point of view, the incremental cost-utility ratio of VNS to treat patients suffering from RD.

DETAILED DESCRIPTION:
Depression is a common illness, affecting 17% of the population over the course of a lifetime. A third of depressions relapses and progresses to recurrence and resistance to treatments. Despite the optimization of antidepressant medical strategies, 20 to 40% of depressions do not respond to treatment. This is particularly worrying as 6% of non-responder patients will die by committing suicide. The term treatment-resistant depression (TRD) is used when two or more (and often many more) well conducted antidepressant treatments from different classes have failed to achieve remission.

Depression has a major impact on quality of life, socio-professional functioning and healthcare consumption. According to the World Health Organization (WHO), depression will be the second cause of healthcare costs in the world by 2020. RD alone accounts for 30 to 40% of the annual cost of depression.

Sometimes, TRD is part of a bipolar illness, a psychiatric condition characterized by the alternation of depressive and maniac episodes that affects 4% of the population. In this case, the challenge is even bigger because (1) antidepressants are no well tolerated, further reducing the therapeutic options in case of resistance, (2) the severity and duration of the depressive episodes are the main factors explaining the deterioration of the quality of life and the increasing cost of cares for these patients. Bipolar RD currently accounts for 20% of all psychiatric spending.

The standard treatment for TRD is electroconvulsive therapy (ECT), which results in a response in 60 to 70% of cases after a few weeks of treatment. However, the improvement is often transient and 40% of patients relapse within 6 months of the initial ECT session. Moreover, ECT is often not well tolerated because of the frequency and the intensity of the memory disorders associated, the repetition of anesthesia and hospitalizations and its social stigma. Refusals and requests to stop ECT are therefore common even when it is effective, as these constraints are sometimes experienced as being unbearable in the long-term. This therapeutic impasse therefore makes TRD a priority public health target to which it is urgent to provide a realistic medico-economical response.

The literature suggests that Vagus Nerve Stimulation (VNS) has unique kinetics of efficacy in depression, particularly in preventing the long-term recurrences, and therefore responding to the lack of effective maintenance treatment in TRD. In fact, the benefits of VNS gradually accumulate over 12-24 months, which makes it complementary to more incisive treatments like ECT. Finally, its efficacy-tolerance profile appears to be similar in uni and bipolar TRD, giving VNS a potentially unique place in the therapeutic arsenal in psychiatry. VNS has been approved for over 15 years as a treatment for RD in the Unites States and Great-Britain.

The hypothesis is that VNS is a medico-economically efficient therapeutic option to overcome the therapeutic impasse in which patients suffering from uni and bipolar DR currently find themselves due to the frequency of relapses under treatment.

The primary objective is to estimate, from a collective point of view, the incremental cost-utility ratio of VNS to treat patients suffering from RD.

The secondary objectives are evaluating the efficacy and the security of the VNS, as well as positioning the VNS in comparison with ECT that is currently the standard treatment for TRD.

This is a national multicenter comparative, open, randomized, controlled, two-parallel group clinical trial evaluating the medico-economic impact of VNS in resistant depression population. Patients (166) suffering from resistant depression will be enrolled over a 24-month period and will be randomized in a (1:1) ratio to receive either Vagus Nerve Stimulation (VNS) along with the Best Medical Treatment (VNS+BMT arm) or the Optimal Medical Treatment only (BMT arm).

Patients meeting all eligibility criteria will be enrolled in the study.

All subjects will be followed by the investigators or designee of the investigator during the whole study period by visits on site.

Number of visits/participant: Both arms will attend: selection visit (VS), inclusion visit (VI) and randomization visit (R), M0, M2, M4, M6, M8, M10, M12, M14, M16, M18, M20, M22 and M24. After the inclusion visit, the experimental arm (VNS + BMT) will further attend a neurosurgical and anesthetic consultation before being hospitalized for the VNS system placement. The patient will finally be hospitalized in psychiatry for about 5 days for switching the device on. If the target intensity has not been reached during this hospitalization, an adjustment visit is planned every month for 6 months in order to progressively increase the stimulation intensity until the target or a therapeutic response. If the target or the therapeutic response is obtained, the settings adjustments rhythm will be at the indiscretion of the psychiatrist. If at the end of the 6 first visits (M1 to M6), the target intensity couldn't be reached or in absence of a satisfying clinical response, a visit will be planned every 3 months (consultation or hospitalization) to keep optimizing the VNS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older ;
* Childbearing women must have an efficient contraception for the whole study period
* Diagnosis of recurrent depressive trouble or persistent depressive disorder or bipolar disorder (according to DSM-5)
* Start of disorder (defined by the occurrence of the first thymus episode: characterized depressive disorder or maniac episode with or without mixed characteristics) for 5 years or more
* At least one of the following criteria:

  * Criterion A: current characterized depressive disorder and characterized depressive disorder for at least 12 months during the last 24 months despite at least four treatments lines at appropriate dosage and duration
  * Criterion B: current treatment by ECT and criteria A before the start of the ECT treatment or ECT dependency criteria
* Patients who, after the nature of the study has been explained to them, have given written consent

Exclusion Criteria:

* Know pregnancy or breastfeeding
* Schizophrenia, schizoaffective disorder or persistent delusional disorder (DSM-5)
* Characterized depressive disorder with psychotic characteristics within 3 months before the inclusion (DSM-5)
* Concomitant participation to another interventional clinical trial, excepted eventual ancillary researches validated by the study scientific committee. Participation to non-interventional researches is allowed.
* Patients receiving enforced cares (ASPDT, ASPPI, ASPDRE, etc.)
* Non-affiliation to a social security regimen or any other social protection regimen
* Disability, according to the investigator, to understand the study or refusal to sign the study consent form (non-francophone patient, cognitive disorders)
* Anticipated disability to attend all the visits, treatments and measures planned by the protocol: severe personality disorder, severe substance addiction, severe intellectual development disorder. In any of those cases, the notion of severity is at the indiscretion of the investigator

Secondary Exclusion Criteria:

* Surgical contraindication to the VNS
* Positive β-HCG (results obtained after the informed consent is signed but before the randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2028-08-26 (Estimated); Study Completion 2030-08-19 (Estimated)

PRIMARY OUTCOMES:
Cost-utility of VNS | Month 24
  Incremental cost-utility ratio of the Vagus Nerve Stimulation (group VNS + optimal medical treatment) in comparison to the control group (optimal medical treatment only) within 24 months of VNS placement

SECONDARY OUTCOMES:
Efficacy of the VNS | Month 24
  Response rate (< 50% amelioration of the QIDS-SR baseline score) cumulative and non-cumulative
Efficacy of the VNS | Month 24
  Remission rate (QIDS-SR score ≤ 5) cumulative and non cumulative
Efficacy of the VNS | Month 24
  CGI (Clinical Global Impression). Three scores: severity of the disease noted out of 7, overall improvement noted out of 7 and therapeutic index noted out of 16.
Efficacy of the VNS | Month 24
  EGF (Functioning Global Evaluation scale). Minimum: 0. Maximum: 100. The higher the score, the higher the level of psychological, social and occupational functioning.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Number of weeks in depression, remission, (hypo)mania and number of major depressive episodes and (hypo)maniac episodes (DSM-5 criteria)
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of anxious symptoms : STAI-A (State-Trait Anxiety Inventory - Form A). Minimum: 20. Maximum: 80. A higher score indicates greater anxiety.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of thymus symptoms : QIDS-SR (Quick Inventory of Depressive Symptomatology - Self Report). Minimum: 0. Maximum: 27. The higher the score, the worse the symptoms.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of thymus symptoms : YMRS (Young Mania Rating Scale). Minimum: 0. Maximum: 60. The higher the score, the more severe the symptoms.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of thymus symptoms : VAS mood (Visual Analogue Scale Mood). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his mood.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of thymus symptoms : VAS motivation (Visual Analogue Scale Motivation). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his motivation.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of depressive episodes : QIDS-SR (Quick Inventory of Depressive Symptomatology - Self Report). Minimum: 0. Maximum: 27. The higher the score, the worse the symptoms.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of depressive episodes : VAS mood (Visual Analogue Scale Mood). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his mood.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of depressive episodes : VAS motivation (Visual Analogue Scale Motivation). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his motivation.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average duration of response periods (< 50% improvement in QIDS-SR baseline score).
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of symptoms during the response phases : QIDS-SR (Quick Inventory of Depressive Symptomatology - Self Report). Minimum: 0. Maximum: 27. The higher the score, the worse the symptoms.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of symptoms during the response phases : VAS mood (Visual Analogue Scale Mood). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his mood.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of symptoms during the response phases : VAS motivation (Visual Analogue Scale Motivation). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his motivation.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of (hypo)maniac episodes: YMRS (Young Mania Rating Scale). Minimum: 0. Maximum: 60. The higher the score, the more severe the symptoms.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of (hypo)manic episodes: VAS mood (Visual Analogue Scale Mood ). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his mood.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average intensity of (hypo)manic episodes: VAS motivation (Visual Analogue Scale Motivation). Cursor to be positioned by the patient on a non-graduated figure in order to reflect his motivation.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average duration of depressive episodes (DSM-5 criteria) and (hypo)manic episodes
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Interval between the major depressive episodes and interval between the (hypo)maniac episodes (DSM-5 criteria)
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Number of treatments/month
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Total cost of cares
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Quality of life : Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire Short Form). Score out of 70 and percentage. The higher the score, the higher the quality of life.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Quality of life : SF-36 (Short Form 36 Health Survey). 8 dimensions each evaluated out of 100. The higher the score, the higher the quality of life.
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Response rate (< 50% improvement in QIDS-C baseline score) cumulative and non-cumulative
Efficacy of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average C-SSRS scoring
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Cumulative number of ECT session within 24 months
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Number of maintenance ECT session within 24 months
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average duration to obtain a complete ECT withdrawal
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Average time period between ECT during the maintenance phase
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Proportion of patients withdraw from ECT
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Number of treatments per year
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Results of EVA memory disorders severity
Impact of the VNS on ECT (electroconvulsive therapy) | Months: 0, 12, 24
  Montreal Cognitive Assessment (MoCA) scoring
Security of the VNS | Months: 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  1/ VNS failure rate with a subgroup analysis for patients concomitantly treated by ECT, 2/Reported serious and non-serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DOMENECH, MD, MSc, Study Director — GHU Paris Psychiatrie & Neurosciences (site Sainte-Anne)
Locations (23):
- France (23):
  - CHU Angers, Angers
  - Centre Hospitalier Charles Perrens, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Hôpital Gabriel Montpied, Clermont-Ferrand
  - AP-HP. Nord - Université de Paris, Hôpital Louis Mourier, Colombes
  - APHP. Hôpitaux Universitaires Henri Mondor, Hôpital Henri Mondor, Créteil
  - CHU Dijon, Hôpital Le Bocage, Dijon
  - CHU Grenoble Alpes, Grenoble
  - AP-HP. Centre - Université de Paris, Hôpital Corentin-Celton, Issy-les-Moulineaux
  - AP-HP. Université Paris Saclay, Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Lille, Lille
  - Hospices Civils de Lyon, Hôpital Pierre Wertheimer, Lyon
  - Assistance Publique Hôpitaux de Marseille, Hôpital de la Conception, Marseille
  - CHU de Nantes, Hôtel Dieu, Nantes
  - CHU Nice, Hôpital Pasteur 1, Nice
  - AP-HP. Sorbonne Université, Hôpital La Pitié Salpetrière, Paris
  - GHU Paris Psychiatrie & Neuroscience, site Saint Anne, Paris
  - Centre Hospitalier Henri Laborit, Poitiers
  - Centre Hospitalier Guillaume Regnier, Rennes
  - CHU Rouen, Centre Hospitalier du Rouvray, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Toulouse, Hôpital de Psychiatrie, Toulouse
  - CHRU Tours, Clinique Psychiatrique Universitaire, Tours

IPD SHARING:
Plan to Share IPD: No
Datas are own by Assistance Publique - Hôpitaux de Paris, please contact sponsor for further information.